# The Experiences of Erotic and Sexual Risk of Transgender Men: Exploratory Research Design

NCT05187442

# 1. Research Objective

This study focuses on transgender men (TM) and uses a respondent-driven sampling (RDS) method to recruit participants through surveys, focus groups, and in-depth interviews. In addition, transgender women (TW) and non-binary individuals are also recruited for focus groups and in-depth interviews. We aim to understand the current state of sexual culture, sexual risk, and experiences of abuse among TM in the country to assess future sexual health care needs. This will serve as a crucial reference for developing guidelines for TM sexual health care and promoting gender-friendly healthcare environments.

### 2. Research Methods and Procedures

### (1) Research Design

This study employs an explanatory design within a mixed methods research approach. Initially, a survey will be conducted to collect data on sexual orientation and sexual risk among transgender men (TM). Subsequently, purposive sampling will be used to select willing survey respondents who meet the criteria for participation in focus groups or semi-structured in-depth interviews, providing an in-depth understanding of sexual experiences, sexual risks, and abuse among TM in Taiwan. Additionally, transgender women (TW) and non-binary individuals will be recruited for focus groups or semi-structured in-depth interviews to explore abuse experiences and variations across gender identities. TM participants will be recruited using respondent-driven sampling (RDS), inviting willing individuals and encouraging them to recommend other potential participants to ensure heterogeneity and diversity in the sample. For the qualitative interviews in the second phase, TW and non-binary participants will be recruited via snowball and purposive sampling to serve as a comparative reference for the qualitative and survey findings among TM.

## (2) Online Survey

To understand the sexual experiences and sexual risk profile of TM in Taiwan, data will be collected through an online survey. This method aims to reduce the pressure of disclosure and broaden the geographic reach of recruitment. After quantitative data analysis, a subset of respondents will be selected for in-depth interviews in the second phase to collect qualitative data. The online survey is expected to take 15-20 minutes to complete.

# • Survey Participant Eligibility

- A. Individuals who are or have been transgender men, regardless of whether they have undergone gender-affirming surgery.
- B. Must be at least 20 years old.
- C. Must reside in Taiwan.

### • Research Tools

Participants will complete a survey on sexual experiences and sexual risk among transgender men. The survey will be conducted via Google Forms, and only fully completed forms will be counted as valid samples. The survey consists of five main sections:

- A. Demographic Data
- B. Gender-related Information (Questionnaire on Sexual & Gender)
- C. Sexual Experience and Intimate Relationships (Questionnaire on Intimate Relationship and Sexual Behavior)
- D. Screening History (Experience with STI/HIV/HPV Testing)
- E. Information on Drug Use

### (3) Focus Groups and In-Depth Interviews

Following the first-year survey analysis, which revealed that nearly 60% of TM participants had experienced abuse, the research team selected diverse TM participants based on their experiences with abuse. Additional TW and non-binary individuals were recruited for focus groups or semi-structured in-depth interviews to compare abuse experiences across gender identities

# • Eligibility for Focus Group or In-Depth Interview Participants (TM/TW/Non-binary groups)

- A. Self-identify as TM, TW, or non-binary.
- B. Must be at least 20 years old.
- C. Hold Republic of China nationality and reside in Taiwan.
- D. Willingness to share personal experiences and interact with other research participants.
- E. Proficiency in Chinese and sufficient verbal ability.
- F. Meet the research team's purposive sampling criteria.

# • Focus Group or In-Depth Interview Outline

Based on survey questions and statistical analysis after the survey is completed, the interview guide will be refined. The questions will center on participants' experiences with abuse, sexual relationships, and sexual risk, delving into their life stories.

- A. Basic Personal Information: Age, residence, current relationship status, etc.
- B. Questions on Experiences of Abuse, Sexual Relationships, and Sexual Risk.

### 3. Data Processing and Analysis

After all data have been coded and recorded, quantitative data will be processed and analyzed using SPSS version 27.0 software. Descriptive statistics, along with Chi-square or Fisher's

Exact test analyses, will be applied. Explanations will be developed based on the findings from the qualitative data analysis to interpret the current conditions. The qualitative data analysis will focus on the content from the in-depth interviews.